CLINICAL TRIAL: NCT05250271
Title: Forecasting and Preventing Post-Bariatric Hypoglycaemia (Work Package 2)
Brief Title: Forecasting and Preventing Post-Bariatric Hypoglycaemia WP 2
Acronym: PBH Forecast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lia Bally (Other)
Collaborators: University of Padova (Other)
Responsible Party: Sponsor-Investigator, Lia Bally, Head of Nutrition, Metabolism and Obesity and Head of Research, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: PBH Forecast (WP 2)
Record Dates: First submitted 2022-01-14; First posted 2022-02-22 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Post-bariatric Hypoglycaemia; Roux-en-Y Gastric Bypass
Keywords: Continuous Glucose Monitoring
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Intervention Model Description: 3-period crossover design
Who Masked: Participant
Masking Description: Participants are blinded to sensor and plasma glucose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment sequence 1 (Other): Sequence of the treatments: Glucose (15g) - Glucose (5g) -Protein bar
  Interventions: Other: 15 g dextrose; Other: 5 g dextrose; Other: Protein bar
- Treatment sequence 2 (Other): Sequence of the treatments: Glucose (15g) - Protein bar - Glucose (5g)
  Interventions: Other: 15 g dextrose; Other: 5 g dextrose; Other: Protein bar
- Treatment sequence 3 (Other): Sequence of the treatments: Glucose (5g) - Glucose (15g) - Protein bar
  Interventions: Other: 15 g dextrose; Other: 5 g dextrose; Other: Protein bar
- Treatment sequence 4 (Other): Sequence of the treatments: Glucose (5g) - Protein bar - Glucose (15g)
  Interventions: Other: 15 g dextrose; Other: 5 g dextrose; Other: Protein bar
- Treatment sequence 5 (Other): Sequence of the treatments: Protein bar - Glucose (15g) - Glucose (5g)
  Interventions: Other: 15 g dextrose; Other: 5 g dextrose; Other: Protein bar
- Treatment sequence 6 (Other): Sequence of the treatments: Protein bar - Glucose (5g) - Glucose (15g)
  Interventions: Other: 15 g dextrose; Other: 5 g dextrose; Other: Protein bar

INTERVENTIONS:
Other: 15 g dextrose — 15 g dextrose tablets
Other: 5 g dextrose — 5 g dextrose tablets
Other: Protein bar — 5 g carbohydrates + 10 g protein

SUMMARY:
The overall aim of this study is to develop a sustainable hypoglycemia correction strategy.

DETAILED DESCRIPTION:
Obesity is a major global public health concern, for which the most effective therapy is bariatric surgery. Beyond weight loss, bariatric surgery exerts powerful effects on glucose metabolism, achieving complete type 2 diabetes remission in up to 70% of cases. An exaggeration of these effects, however, can result in an increasingly recognized metabolic complication known as postprandial hyperinsulinaemic hypoglycaemia or post-bariatric hypoglycaemia (PBH). The condition manifests 1-3 years after surgery with meal-induced hypoglycaemic episodes. Emerging data suggests that PBH is more frequent than previously thought and affects approximately 30% of postoperative patients, more commonly after gastric bypass than sleeve gastrectomy. Of note, asymptomatic PBH is common, as shown in studies using continuous glucose monitoring (CGM). It is known from extensive research in people with diabetes that recurrent episodes of hypoglycaemia impair counter regulatory defences against subsequent events, predisposing patients to severe hypoglycaemia.

Despite the increasing prevalence of PBH, clinical implications in this population are still unclear. Anecdotal evidence from patients with PBH suggests a high burden for these patients due to the recurrent hypoglycaemias with possibly debilitating consequences. It is well established that even mild hypoglycaemia (plasma glucose of 3.4 mmol/L) in diabetic and non-diabetic patients impairs various cognitive domains. Of note, some of the cognitive functions remain impaired for up to 75 min, even when the hypoglycaemia is corrected. Further concerns exist from observational studies showing associations between PBH during pregnancy and poor foetal growth.

Thus, it is important to timely detect and treat hypoglycaemia with an intervention that allows quick recovery of glycaemia to a safe level, thereby alleviating symptoms and eliminating the risk of potentially hazardous sequelae. Current diabetes-inspired guidelines recommend to correct hypoglycaemia with 15-20 g fast-acting carbohydrates, preferably glucose. However, clinical experience with PBH patients shows that the rapid spikes in glycaemia following correction of hypoglycaemia with such proposed strategies may trigger rebound hypoglycaemia in PBH patients. However, hypoglycaemia correction strategies that are tailored to the specific needs of PBH do not exist currently. Previous research suggests that glucose co-ingested with amino acids induces a metabolic environment that could be favourable for PBH patients due to elevated glucagon levels. However, it currently remains speculative whether combinations of amino acids with glucose could offer more suitable and sustainable PBH correction strategies.

Given the potentially hazardous consequences of hypoglycaemia, development of hypoglycaemia management strategies to adequately predict and treat critical blood glucose levels in the PBH population are urgently needed. Such strategies have to significantly lower the burden of PBH and increase patient safety.

The overall aim or the PBH forecast project (containing 3 WPs) is to prevent hypoglycaemic events in patients with PBH and to develop a sustainable hypoglycaemia correction strategy. The primary objective of WP 2 is to test different nutritional strategies for sustainable hypoglycaemia correction (e.g. minimising time spent hypoglycaemic without causing rebound hyper- and hypoglycaemia).

ELIGIBILITY:
Inclusion Criteria:

* Post-bariatric surgery patients (Roux-en-Y gastric bypass) with PBH, defined as postprandial plasma or sensor glucose <3.0 mmol/L according to the International Hypoglycaemia Study Group and exclusion of other causes of hypoglycaemia
* Age ≥18 years

Exclusion Criteria:

* Inability to give informed consent as documented by signature
* Pregnant or lactating women
* Inability or contraindications to undergo the investigated intervention
* Drugs interfering with blood glucose (e.g. SGLT-2 inhibitors, acarbose) during the time of investigation
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Time in glucose target range | During 40 minutes after hypoglycaemia correction
  The primary endpoint is time in glucose target range (plasma glucose 3.9-5.5 mmol/L).

SECONDARY OUTCOMES:
Percentage of time with plasma glucose <3.0 mmol/L | During 40 minutes after hypoglycaemia correction
  Units: %
Percentage of time with plasma glucose <3.9 mmol/L | During 40 minutes after hypoglycaemia correction
  Units: %
Percentage of time with plasma glucose >5.5 mmol/L | During 40 minutes after hypoglycaemia correction
  Units: %
Percentage of time with plasma glucose >10.0 mmol/L | During 40 minutes after hypoglycaemia correction
  Units: %
Percentage of time with sensor glucose <3.0 mmol/L | During 150 minutes after hypoglycaemia correction
  The sensor glucose values will be adjusted to plasma glucose to increase accuracy
Percentage of time with sensor glucose <3.9 mmol/L | During 150 minutes after hypoglycaemia correction
  The sensor glucose values will be adjusted to plasma glucose to increase accuracy
Percentage of time with sensor glucose >5.5 mmol/L | During 150 minutes after hypoglycaemia correction
  The sensor glucose values will be adjusted to plasma glucose to increase accuracy
Percentage of time with sensor glucose >10.0 mmol/L | During 150 minutes after hypoglycaemia correction
  The sensor glucose values will be adjusted to plasma glucose to increase accuracy
Peak plasma glucose | Until 40 minutes after inital hypoglycaemia correction or 180 minutes after meal intake (the later timepoint of the two)
  Peak plasma glucose (mmol/L)
Time to euglycaemia | Until 40 minutes after inital hypoglycaemia correction or 180 minutes after meal intake (the later timepoint of the two)
  Time to euglycaemia after hypoglycaemia correction (plasma glucose ≥3.9 mmol/L)
Rebound hypoglycaemia | During 150 minutes after hypoglycaemia correction
  Proportion of participants with rebound hypoglycaemia (plasma glucose <3.0 mmol/L following successful primary hypoglycaemia correction defined as plasma glucose ≥3.9 mmol/L)
Insulin | 15 minutes after hypoglycaemia correction
  Serum insulin concentration
Glucagon | 15 minutes after hypoglycaemia correction
  Serum glucagon concentration

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, Prof. Dr. med. et phil., Principal Investigator — Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, lnselspital, Bern University Hospital, University of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism (UDEM), Inselspital, Bern University Hospital, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available to other researchers.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After study completion, 10 years
Access Criteria: Data will be shared after written inquiry and approval by the principal investigator.